CLINICAL TRIAL: NCT04432298
Title: Randomized, Double-Blind, Placebo-Controlled Phase 2 Study of the Efficacy and Safety of Intravenous Pamrevlumab, a Monoclonal Antibody Against Connective Tissue Growth Factor (CTGF), in Hospitalized Patients With Acute COVID-19 Disease
Brief Title: Study of the Efficacy and Safety of Intravenous Pamrevlumab, in Hospitalized Participants With Acute COVID-19 Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated by Sponsor due to low enrollment.
Sponsor: Kyntra Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FGCL-3019-098
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Results first posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-06

CONDITIONS: COVID-19
Keywords: Severe Acute Respiratory Syndrome coronavirus; SARS-COV-2 infection
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome | interventions — pamrevlumab

STUDY DESIGN:
Intervention Model Description: Proof-of-concept
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pamrevlumab (Experimental): Pamrevlumab: 35 milligrams/kilogram (mg/kg) on Days 1, 7, 14 and 28 for a total of 4 infusions over 4 weeks
  Interventions: Drug: Pamrevlumab
- Placebo (Experimental): Pamrevlumab-matching placebo on Days 1, 7, 14 and 28 for a total of 4 infusions over 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pamrevlumab — Sterile liquid for injection
  Other Names: FG-3019
  Arms: Pamrevlumab
Drug: Placebo — Sterile liquid for injection
  Arms: Placebo

SUMMARY:
This study evaluates the efficacy and safety of intravenous (IV) infusions of pamrevlumab when compared with placebo in participants who are hospitalized with acute COVID-19 disease.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, phase 2, proof-of-concept study to evaluate the efficacy and safety of IV pamrevlumab, a monoclonal antibody, against connective-tissue growth factor (CTGF), in participants hospitalized with acute COVID-19 disease.

All concomitant medications, including approved and non-approved treatments for COVID-19 (such as, hydroxychloroquine or interleukin 6 [IL-6] inhibitors), as well as supplemental oxygenation needs, will be collected and recorded. In addition, the following will be collected and recorded: documentation of Severe Acute Respiratory Syndrome coronavirus (SARS-Cov-2) infection, documentation of any other infection(s) prior to or during hospitalization, and whether or not aggressive care is withheld or withdrawn, including the reason for withholding or withdrawal of care (such as a Do Not Resuscitate/Do Not Intubate [DNR/DNI] order or a resource limitation).

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed SARS-CoV-2 infection
2. Respiratory compromise requiring hospitalization for COVID-19 disease as evidenced by at least one (or more) of the following criteria:

   * Interstitial pneumonia on chest x-ray or high-resolution computed tomography (findings of consolidation or ground glass opacities), OR
   * Peripheral capillary oxygen saturation < 94% on room air, OR
   * Requiring non-invasive supplemental oxygen (such as, nasal cannula, face mask) to maintain SpO2
3. Not requiring mechanical ventilation and/or extracorporeal membrane oxygenation (ECMO) use at time of randomization
4. Not participating in another clinical trial for the treatment of COVID-19 disease through Day 28

Exclusion Criteria:

1. Female participants who are pregnant or nursing
2. Participation in a clinical trial with another investigational drug for COVID-19 disease
3. Anticipated discharge from the hospital or transfer to another hospital or long-term care facility which is not a study site within 72 hours of randomization
4. History of allergic or anaphylactic reaction to human, humanized, chimeric or murine monoclonal antibodies

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-06-20 (Actual); Primary Completion 2021-03-22 (Actual); Study Completion 2021-03-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Research Center, Detroit, Michigan
  - Research Center, Greensboro, North Carolina
  - Research Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pamrevlumab | Placebo
Started | 11 | 11
Intent-to-Treat (ITT) Population (All randomized participants) | 11 | 11
Safety Population (Received at least 1 dose of study drug) | 9 | 11
Completed | 5 | 8
Not Completed | 6 | 3
Not completed — Other than specified | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 3 | 2
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: ITT population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pamrevlumab | Placebo | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (10) | 61 (14) | 61 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 7 | 8 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 8
  Not Hispanic or Latino | 5 | 8 | 13
  Unknown or Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2 | 6 | 8
  Black or African American | 3 | 2 | 5
  Other | 5 | 2 | 7
  Unknown | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Alive Who Never Received Mechanical Ventilation and/or Extracorporeal Membrane Oxygenation (ECMO) at Day 28
Time Frame: Day 28
Population: ITT Population: All randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Pamrevlumab | Placebo
Number analyzed (Participants) | 11 | 11
Participants | 8 | 9

2. Secondary Outcome: Number of Participants Alive, Discharged Home, and Not on Supplemental Oxygen at Day 28
Time Frame: Day 28
Population: ITT Population: All randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Pamrevlumab | Placebo
Number analyzed (Participants) | 11 | 11
Participants | 6 | 7

3. Secondary Outcome: Number of Participants Alive Who Never Received Mechanical Ventilation and/or ECMO at Day 14
Time Frame: Day 14
Population: ITT Population: All randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Pamrevlumab | Placebo
Number analyzed (Participants) | 11 | 11
Participants | 8 | 9

4. Secondary Outcome: Time to Recovery as Based on a Modified 8-Point Ordinal Scale
Description: Recovery was defined as the first day on which the participant satisfied 1 of the following 3 categories from the 8-point ordinal scale: (1) hospitalized, not requiring supplemental oxygen; (2) Not hospitalized (discharged), but with limitation on activities and/or requiring home supplemental oxygen; (3) Not hospitalized (discharged), with no limitations on activities and not requiring supplemental oxygen).
Time Frame: Day 28
Population: ITT Population: All randomized participants. Here, overall number of participants analyzed signifies those who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Pamrevlumab | Placebo
Number analyzed (Participants) | 6 | 8
days | 11 (10) | 11 (12)

5. Secondary Outcome: Days in Intensive Care Unit/Critical Care Unit (ICU/CCU) (Either on or Off Mechanical Ventilation and/or ECMO)
Description: Days in ICU/CCU was calculated as Event end date/time - Event start data/time + 1. Participants who died in ICU/CCU before Day 28, days in ICU/CCU is calculated up to the death date. Days in ICU/CCU were censored after Day 28.
Time Frame: up to Day 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Pamrevlumab | Placebo
Number analyzed (Participants) | 4 | 3
days | 16 (14) | 12 (17)

6. Secondary Outcome: Days on Mechanical Ventilation and/or ECMO
Description: Days on Mechanical Ventilation and/or ECMO was calculated as Event end date/time - Event start data/time. Participants who died on MV/ECMO before Day 28, days on MV/ECMO is calculated up to the death date. Days on MV/ECMO are censored after Day 28.
Time Frame: up to Day 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Pamrevlumab | Placebo
Number analyzed (Participants) | 2 | 2
days | 20.5 (0.0) | 8.7 (11.1)

7. Secondary Outcome: Time to Mechanical Ventilation/ECMO or All-cause Mortality
Description: Time (number of days) from randomization to mechanical ventilation/ECMO or all-cause mortality by Day 28. Participants without the event are not included in the calculation.
Time Frame: up to Day 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Pamrevlumab | Placebo
Number analyzed (Participants) | 3 | 2
days | 14 (11) | 14 (1)

8. Secondary Outcome: Number of Participants With All-cause Mortality
Time Frame: up to Day 28
Population: ITT Population: All randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Pamrevlumab | Placebo
Number analyzed (Participants) | 11 | 11
Participants | 2 | 1

9. Secondary Outcome: Changes in Pressure of Arterial Oxygen to Fractional Inspired Oxygen Concentration (PaO2/FiO2) Ratio, Both as Categorical and Continuous Variables
Time Frame: up to Day 28
Population: Due to early termination of the study, data was not collected for the assessment.
Arm/Group | Pamrevlumab | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Time to Death From Any Cause
Description: Time (number of days) from randomization to death from any cause by Day 28. Participants without the event are not included in the calculation.
Time Frame: up to Day 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Pamrevlumab | Placebo
Number analyzed (Participants) | 2 | 1
days | 17 (15) | 13 (NA) — Not evaluable due to small number of events.

11. Secondary Outcome: Change in Resting Peripheral Oxygen Saturation (SpO2) Adjusted by FiO2
Time Frame: up to Day 28
Population: Due to early termination of the study, data was not collected for the assessment.
Arm/Group | Pamrevlumab | Placebo
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Change in (Non-invasive) Oxygen Supplementation Requirements
Time Frame: up to Day 28
Population: Due to early termination of the study, data was not collected for the assessment.
Arm/Group | Pamrevlumab | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Day 28
Description: Serious and Other (Not Including Serious) Adverse Events were monitored/assessed for the Safety Population and All-Cause Mortality was monitored/assessed for ITT Population. The ITT Population included all randomized participants. The Safety Population included all participants who received at least 1 dose of study drug. Two participants in the Pamrevlumab group did not receive study drug and were not included in the Safety Population.
Arm/Group | Pamrevlumab | Placebo
All-Cause Mortality (participants affected / at risk) | 3/11 | 2/11
Serious Adverse Events (participants affected / at risk) | 5/9 | 2/11
Other Adverse Events (participants affected / at risk) | 4/9 | 8/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pamrevlumab (N=9) | Placebo (N=11)
Angina pectoris (Cardiac disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Shock (Vascular disorders) | 1 | 1
Peripheral artery thrombosis (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pamrevlumab (N=9) | Placebo (N=11)
Leukocytosis (Blood and lymphatic system disorders) | 2 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Polycythaemia (Blood and lymphatic system disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Adrenal mass (Endocrine disorders) | 1 | 0
Vision blurred (Eye disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Platelet count decreased (Investigations) | 0 | 2
Transaminases increased (Investigations) | 1 | 1
Blood glucose increased (Investigations) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Due to early termination of this study, formal analyses of the primary and secondary endpoints are not presented because the study's sample size is substantially underpowered for meaningful interpretation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The multisite consortium can publish any time after the data is collected and analyzed by FibroGen. The investigator can only publish after the multisite consortium publishes (or tries to publish and fails). FibroGen has 60 days to review a publication and can extend the embargo up to an additional 120 days (or 180 total).

DOCUMENTS (2):
  • Study Protocol (2020-05-12): https://cdn.clinicaltrials.gov/large-docs/98/NCT04432298/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/98/NCT04432298/SAP_001.pdf